CLINICAL TRIAL: NCT03364205
Title: The Effect of the Solution Focused Approach (SFA) on Nutrition-Exercise Attitudes and Behaviors of Overweight and Obese Adolescents: Randomized Controlled Trial
Brief Title: Solution Focused Approach in Adolescents (SFA)
Acronym: SFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Nurcan AKGUL-GUNDOGDU, Assistant Professor, Cumhuriyet University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CumhuriyetU
Record Dates: First submitted 2017-11-14; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Obesity; Overweight and Obesity; Adolescent Obesity
Keywords: SFA interview technique; adolescence; obesity; nutrition; exercise
MeSH Terms: conditions — Obesity; Overweight; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trials
Who Masked: Investigator
Masking Description: There was no intervention in the control group which was in parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): solution-focused interview techniques
  Interventions: Behavioral: solution-focused interview technique
- control (No Intervention): This group did not apply solution-focused interview techniques.

INTERVENTIONS:
Behavioral: solution-focused interview technique — This approach helps an individual make decisions about behavioral change, focusing particularly on his or her past achievements and looking forward to a time when the problems cease to exist.
  Arms: intervention

SUMMARY:
Aims-objectives: This study assessed the effect of the Solution Focused Approach (SFA) interview technique on overweight/obese adolescents' nutrition-exercise attitudes and behaviors.

Background: Obesity is a serious health problem for all age groups, particularly adolescents; therefore, it is important for adolescents to develop healthy nutrition habits, acquire exercise behaviors. Unless healthy nutrition-exercise behaviors are acquired, obesity can develop in adolescence, continue in adulthood. Focusing on solutions can be effective for overweight/obese adolescents to develop healthy nutrition-exercise behaviors.

Design: A pretest-posttest randomized-controlled trial design was used.

Methods: The study included 32 overweight/obese adolescents (16 for intervention group, 16 for control group) aged12-13 years who attended a health center, met the inclusion criteria. The SFA interview technique was applied to the intervention group. Eight solution-focused interviews were conducted with each adolescent at two-week intervals (interview length 30 to 45minutes). For each group, anthropometric, metabolic measurement follow-ups were conducted in the first and sixth months. The data were evaluated using independent samples t-test, Mann-Whitney U, Wilcoxon test respectively for normally, non-normally distributed variables. The categorical variables were compared using chi-square test. The value p<0.05 was accepted to be statistically significant.

DETAILED DESCRIPTION:
Solution Focused Approach (SFA) interview technique is an approach that can be used by nurses who have important roles in the protection, maintenance and promotion of health in healthcare services. Because the SFA interview technique can be integrated into all dimensions of health, it enables children and adolescents to be aware of their own strengths and skills and to improve their skills. This raised awareness encourages individuals to start and maintain change. The earlier the awareness of individuals is raised, the higher the achievement level of the approach will increase. Further studies can be conducted in which the duration of the SFA interview technique follow-ups is longer. Moreover, it can be suggested that studies be conducted to analyze the cost-effectiveness of this approach.

All health professionals in general and, specifically nurses, should be educated about the SFA interview technique strategies. Nurses who carry out the SFA interviews conducted using the SFA interview technique should enable individuals to realize their own strengths. The number of interviews can be determined in accordance with the topic and the data obtained from individuals. If the interviews are carried out with school children-adolescents, attention should be paid to conduct interviews with their families. Enabling individuals to reach a solution using the SFA interview technique strategies is the major point of interviews. This result may not appear immediately. Interviews should be continued with patience to find what works in resistant individuals.

After these interviews are completed, interviews should be continued with the individuals periodically. To enable individuals to maintain their nutrition and exercise behaviors, interviews should be carried out with adolescents and their families at least twice in a month after the SFA interviews. Nurses who conduct SFA interviews can carry out individual interviews or group interviews in Endocrinology Polyclinics, Family Health Centers, or at schools as a school nurse.

ELIGIBILITY:
Inclusion Criteria:

* Twelve-thirteen aged between,
* Diagnosed metabolic disease, without
* BMI >85 percentile (>+1SD), overweight and BMI>95 (>+2SD) percentile obese adolescents
* Communicate
* Any conditions that interfere with exercise (who do not have disability, such as cardiac failure)

Exclusion Criteria:

* From teenagers who indicated they could not continue until the end of the study,
* Metabolic disease,
* Metformin uses
* Adolescents who move out of County

Ages: 12 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2013-09-02 (Actual); Primary Completion 2014-01-29 (Actual); Study Completion 2014-08-29 (Actual)

PRIMARY OUTCOMES:
the Family and Adolescent Introductory Information Form and Overweight and Obese Adolescents' Nutrition-Exercise Behavior Identification Form | one month
  The data for the nutrition-exercise habits and behaviors of the adolescent were collected using the Family and Adolescent Introductory Information Form and Overweight-Obese Adolescents' Nutrition-Exercise Behavior Identification Form, which had been prepared by the researcher based on the literature.
Anthropometric measurement (weight measurement) | one month
  Anthropometric scores (weight measurement) data of adolescents were collected using the Anthropometric Follow-Up Table. Digital weighing scale was used for weight measurements in kilograms. The measurements were taken without closes and shoes. Calibration of the scales was done monthly. The primary outcome was to determine weight measurement values of adolescent.
Anthropometric measurement (height measurement) | one month
  Anthropometric scores (height measurement) data of adolescents were collected using the Anthropometric Follow-Up Table. Bar scale was used for height measurements in meters. Before the length measurement, the shoe was removed and the lower end of the rod was attached to the foot in a vertical position, and the point where the head came was recorded. The primary outcome was to determine height measurement values of adolescent.
Anthropometric measurement (Calculation of Body Mass Index or BMI) | one month
  BMI was calculated as the body mass in kilograms divided by the square of the body height in meters (BMI = kg / m ^ 2). The primary outcome was to determine BMI values of adolescent.
Anthropometric measurement (Body Mass Index Percentile (BMI percentile) calculation) | one month
  In determining the BMI percentile standard values, the BMI values determined for Turkish children were taken into consideration. The primary outcome was to determine BMI percentile values of adolescent.
Anthropometric measurement (Body Mass Index - Standard Deviation Score(BMI-SDS) calculation) | one month
  The data on the Anthropometric scores (BMI-SDS) of the adolescents were collected using the Anthropometric Follow-Up Table. The obtained SDS value is calculated by using the Auxology program which performs SDS calculation.The primary outcome was to determine BMI-SDS values of adolescent.
Metabolic measurement (Preprandial Blood Glucose) | one month
  The data on the Metabolic scores (Preprandial Blood Glucose) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The primary outcome was to determine Preprandial Blood Glucose values of adolescent.
Metabolic measurement (Preprandial insulin) | one month
  The data on the Metabolic scores (Preprandial insulin) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The primary outcome was to determine Preprandial insulin values of adolescent.
Metabolic measurement (Homeostasis Model of Assesment for insulin Resistance (HOMA-IR)) | one month
  The data on the Metabolic scores (Homeostasis Model of Assesment for insulin Resistance (HOMA-IR)) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The primary outcome was to determine HOMA-IR values of adolescent.
Metabolic measurement (LDL-cholesterol) | one month
  The data on the Metabolic scores (LDL-cholesterol) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The primary outcome was to determine LDL-cholesterol values of adolescent.
Metabolic measurement (HDL-cholesterol) | one month
  The data on the Metabolic scores (HDL-cholesterol) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The primary outcome was to determine HDL-cholesterol values of adolescent.
Metabolic measurement (Total cholesterol) | one month
  The data on the Metabolic scores (total cholesterol) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The primary outcome was to determine total cholesterol values of adolescent.
Metabolic measurement (Triglyceride) | one month
  The data on the Metabolic scores (triglyceride) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The primary outcome was to determine triglyceride values of adolescent.
the application of scale - Nutrition-Exercise Attitude Scale (NEAS) | one month
  Healthy nutrition-exercise attitudes and behaviors were evaluated using the Nutrition-Exercise Attitude Scale (NEAS) that had been developed to determine the attitudes and behaviors of the adolescents.The NEAS scores ranged from 13 to 65. A high total score obtained in this scale indicated a positive nutrition-exercise attitude and a low total score indicated a negative attitude.These scales were completed in the first-month follow-up.
the application of scale - Nutrition-Exercise Behavior Scale (NEBS) | one month
  Healthy nutrition-exercise attitudes and behaviors were evaluated using the Nutrition-Exercise Behavior Scale (NEBS) that had been developed to determine the attitudes and behaviors of the adolescents.The NEBS had the following sub-scales: psychological (dependent) eating behavior (11 to 55 points), healthy nutrition-exercise behavior (14 to 70 points), unhealthy nutrition-exercise behavior (14 to 70 points) and regular meal times (6 to 30 points). A high total score obtained in this scale indicated a positive nutrition-exercise behavior and a low total score indicated a negative behavior.These scales were completed in the first-month follow-up.

SECONDARY OUTCOMES:
Anthropometric measurement (weight measurement) | six month
  Anthropometric scores (weight measurement) data of adolescents were collected using the Anthropometric Follow-Up Table. Digital weighing scale was used for weight measurements in kilograms. The measurements were taken without closes and shoes. Calibration of the scales was done monthly. The second outcome was to enable the weight measurement values to be within the reasonable limits.
Anthropometric measurement (height measurement) | six month
  Anthropometric scores (height measurement) data of adolescents were collected using the Anthropometric Follow-Up Table. Bar scale was used for height measurements in meters. Before the length measurement, the shoe was removed and the lower end of the rod was attached to the foot in a vertical position, and the point where the head came was recorded. The second outcome was to enable the height measurement values to be within the reasonable limits.
Anthropometric measurement (Calculation of Body Mass Index or BMI) | six month
  BMI was calculated as the body mass in kilograms divided by the square of the body height in meters (BMI = kg / m ^ 2). The second outcome was to enable the BMI values to be within the reasonable limits.
Anthropometric measurement (Body Mass Index Percentile (BMI percentile) calculation) | six month
  In determining the BMI percentile standard values, the BMI values determined for Turkish children were taken into consideration. The second outcome was to enable the BMI percentile values to be within the reasonable limits.
Anthropometric measurement (Body Mass Index - Standard Deviation Score(BMI-SDS) calculation) | six month
  The data on the Anthropometric scores (BMI-SDS) of the adolescents were collected using the Anthropometric Follow-Up Table. The obtained SDS value is calculated by using the Auxology program which performs SDS calculation. The second outcome was to enable the BMI-SDS values to be within the reasonable limits.
Metabolic measurement (Preprandial Blood Glucose) | six month
  The data on the Metabolic scores (Preprandial Blood Glucose) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The second outcome was to enable the Preprandial Blood Glucose values to be within the reasonable limits.
Metabolic measurement (Preprandial insulin) | six month
  The data on the Metabolic scores (Preprandial insulin) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The second outcome was to enable the Preprandial insulin values to be within the reasonable limits.
Metabolic measurement (Homeostasis Model of Assesment for insulin Resistance (HOMA-IR)) | six month
  The data on the Metabolic scores (HOMA-IR) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The second outcome was to enable the HOMA-IR values to be within the reasonable limits.
Metabolic measurement (LDL-cholesterol) | six month
  The data on the Metabolic scores (LDL-cholesterol) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The second outcome was to enable the LDL-cholesterol values to be within the reasonable limits.
Metabolic measurement (HDL-cholesterol) | six month
  The data on the Metabolic scores (HDL-cholesterol) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The second outcome was to enable the HDL-cholesterol values to be within the reasonable limits.
Metabolic measurement (Total cholesterol) | six month
  The data on the Metabolic scores (total cholesterol) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The second outcome was to enable the total cholesterol values to be within the reasonable limits.
Metabolic measurement (Triglyceride) | six month
  The data on the Metabolic scores (triglyceride) of the adolescents were collected using the Metabolic Follow-Up Table.These tables were completed by both groups before the first- and sixth- follow-ups between September 6 2013 and August 29 2014. The second outcome was to enable the triglyceride values to be within the reasonable limits.
the application of scale- Nutrition-Exercise Attitude Scale (NEAS) | six month
  Healthy nutrition-exercise attitudes and behaviors were evaluated using the Nutrition-Exercise Attitude Scale (NEAS) that had been developed to determine the attitudes and behaviors of the adolescents.The NEAS scores ranged from 13 to 65. A high total score obtained in this scale indicated a positive nutrition-exercise attitude and a low total score indicated a negative attitude.These scales were completed in the sixth-month follow-up.
the application of scale - Nutrition-Exercise Behavior Scale (NEBS) | six month
  Healthy nutrition-exercise attitudes and behaviors were evaluated using the Nutrition-Exercise Behavior Scale (NEBS) that had been developed to determine the attitudes and behaviors of the adolescents.The NEBS had the following sub-scales: psychological (dependent) eating behavior (11 to 55 points), healthy nutrition-exercise behavior (14 to 70 points), unhealthy nutrition-exercise behavior (14 to 70 points) and regular meal times (6 to 30 points). A high total score obtained in this scale indicated a positive nutrition-exercise behavior and a low total score indicated a negative behavior.These scales were completed in the sixth-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Emine- Ümit SEVİG, 2, Study Director — TC Erciyes University; Nuran Güler, 3, Study Director — Cumhuriyet University
Locations (1):
- Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Journal of Clinical Nursing
Supporting Information: Analytic Code
Time Frame: Until 2018
Access Criteria: For editorial review
URL: http://onbehalfof+jcn+wiley.com@manuscriptcentral.com